CLINICAL TRIAL: NCT05815472
Title: Advanced Patient Monitoring and A.I. Supported Outcomes Assessment in Lung Cancer Using Internet of Things Technologies (A.I. - APALITT)
Acronym: APALITT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3817
Record Dates: First submitted 2023-03-13; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients affected by locally advanced non-small-cell lung cancer (Experimental): Patients affected by locally advanced non-small-cell lung cancer (staged III according to 8th TNM classification), undergoing induction therapy (IT) followed by either radical surgery or immunotherapy boost and treated in Fondazione Policlinico Universitario "A. Gemelli" IRCCS of Rome, Italy, will be enrolled in this study.
  Interventions: Device: Fitbit charge

INTERVENTIONS:
Device: Fitbit charge — Internet of Things Technologies Device

SUMMARY:
The use of advanced technological tools able to exploit patient-centered "Real World Data", represents an innovative and fascinating challenge for the most modern personalized medicine paradigms.

Monitoring oncological patients during multimodal cancer therapies may represent a significant step towards a comprehensive and reliable quality of life assessment, prevention of toxicity before its clinical onset and treatment outcomes prediction.

The big data approach, being able to collect, manage and interpret large volumes of health data, eventually supported by artificial intelligence (A.I.) is therefore fundamental in this setting and may be translated in the next future in tangible advantages for the patients.

Primary aim of the project is to assess patients experience of using portable monitoring systems during multimodal oncological therapies and follow up period, through the use of a dedicated app and wearable technology (i.e. monitoring bracelet), as Electronic Health Record data harvesting devices.

More specifically, the patients report experience measure of man/women affected by locally advanced non-small-cell lung cancer undergoing chemo(radio)therapy followed either by surgery or immunotehrapy (e.g. describing toxicity, instrumental activities of daily living and stress/coping levels) will be analyzed.

The machine learning assisted analysis of these data will allow to identify patients profile that may be used as risk categories to optimize assistance and follow up practices.

This is an observational study with device, co-financed, monocentric study with a foreseen study duration of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged < 75
* Clinically able to use portable technologies
* Able to understand and sign informed consent

Exclusion Criteria:

* Major psychiatric disorder
* ECOG>2 performance status
* Not able to use portable technologies

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-09-28 (Estimated)

PRIMARY OUTCOMES:
Daily collection of basis real world data such as physical activity in non-small-cell lung cancer patients by portable monitoring systems | 8-52 weeks
  Patients will receive a state-of -the-art wearable device (electronic wrist bracelet) that will collect real world data everyday such as physical activity that will be established on the basis of the number of steps per day.
  The device will be delivered to patients during the first appointment prior to the beginning of chemotherapy and/or radiotherapy. The collected data will be then transferred to the patient's paired device through the application Healthentia downloaded on appropriate instruments (e.g. smartphone). Data will be collected during multimodal oncological therapies and follow-up period.
Daily collection of basis real world data such as sleep habits in non-small-cell lung cancer patients by portable monitoring systems | 8-52 weeks
  Patients will receive a state-of -the-art wearable device (electronic wrist bracelet) that will collect real world data everyday such as sleep habits that will be established on the basis of the number of sleeping hours.
Daily collection of basis real world data such as vital signs in non-small-cell lung cancer patients by portable monitoring systems | 8-52 weeks
  Patients will receive a state-of -the-art wearable device (electronic wrist bracelet) that will collect real world data everyday such as vital signs that will be established on the basis of heartbeats per minute. A normal resting heart rate should be between 60 to 100 beats per minute.

SECONDARY OUTCOMES:
The completion of Lawton Instrumental Activities of Daily Living questionnaire | 8-52 weeks
  During the whole observation period, patients will be also asked to report their independent living skills through the same application, completing the dedicated questionnaire with the following scoring systems. The Lawton Instrumental Activities of Daily Living (IADL) will be evaluated using the Lawton Brody instrumental scale. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and from 0 to 5 for men (8-items version).
The completion of the EORTC QLQ-C30 questionnaire | 8-52 weeks
  During the whole observation period, patients will be also asked to report their Quality of Life through the same application, completing the dedicated questionnaire with the following scoring systems. The EORTC QLQ-C30 questionnaire comprises 30 items, 24 of which are combined into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnea, sleep disorders, appetite loss, diarrhea, constipation, and the financial impact) scales assess symptoms. All of the scales and single-item measures range in score from 0 to 100. Higher score for global health status and functioning scales indicates a better level of functioning, whereas higher scores on symptom-oriented scales means more severe symptoms.
The completion of the Malnutrition Screening Tool | 8-52 weeks
  During the whole observation period, patients will be also asked to report their nutritional status through the same application, completing the dedicated questionnaire with the following scoring systems. The Malnutrition Screening Tool is an easy two question screening tool that evaluates the level of malnutrition risk, giving a score out of five.
  To calculate the total score, add the point(s) from question one and question two together to get a total.
  * A score of 0 - 1 indicates a low risk of malnutrition.
  * A score of 2 indicates a moderate risk of malnutrition.
  * A score of 3 - 5 indicates a high risk of malnutrition.
The completion of the Distress thermometer - DT6 test | 8-52 weeks
  During the whole observation period, patients will be also asked to report their psychological status through the same application, completing the dedicated questionnaire with the following scoring systems. The distress thermometer (DT) is an efficient tool for identifying distress among cancer patients worldwide. The National Comprehensive Cancer network (NCCN) Distress Thermometer (DT) is a one-item, 11-point Likert scale depicted as a visual graphic of a thermometer that ranges from 0 (no distress) to 10 (extreme distress), with which patients indicate their level of distress over the course of the week prior to assessment.
The completion of Mental Adjustment to Cancer Scale - MINI-MAC 7 questionnaire | 8-52 weeks
  During the whole observation period, patients will be also asked to report their psychological status through the same application, completing the dedicated questionnaire with the following scoring systems. The Mental Adjustment to Cancer Scale - MINI-MAC 7, Italian version, consists of 29 statements, which aim at measuring four ways of facing cancer, such as Anxiety, Fighting spirit, Helplessness-hopelessness, and Positive reevaluation. Each statement is rated on a scale of 1 (definitely not) to 4 (definitely yes). According to the answers, each of the four ways of dealing with the disease will be rated from 7 to 28 points. The higher the score, the greater the severity of the behaviors in the patient's struggle with cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy